CLINICAL TRIAL: NCT01318265
Title: A Phase I, Non-Randomized, Open Label Study to Determine the Effetc of Ketoconazole on the Pharmacokinetics of a Single Oral Dose of Regorafenib (BAY73-4506) in Healthy Volunteers
Brief Title: Effect of Ketoconazole on Regorafenib (BAY73-4506) Pharmacokinetics
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None
Other Study IDs: 12435
Record Dates: First submitted 2011-02-18; First posted 2011-03-18 (Estimated); Last update posted 2014-11-03 (Estimated); Status verified 2014-10

CONDITIONS: Pharmacokinetics
Keywords: drug interactions; ketoconazole; pharmacokinetics; human volunteers
MeSH Terms: interventions — regorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm1 (Experimental)
  Interventions: Drug: Regorafenib (BAY73-4506); Regorafenib (BAY73-4506) plus ketoconazole

INTERVENTIONS:
Drug: Regorafenib (BAY73-4506); Regorafenib (BAY73-4506) plus ketoconazole — Treatment 1: A single 160 mg dose of BAY73-4506. Treatment 2: Ketoconazole 400 mg once daily from Day -4 to Day 3. A single 160 mg dose of BAY73-4506 on Day 1.

SUMMARY:
The purpose of this study is to estimate the effect of multiple doses of ketoconazole on the pharmacokinetics of a single dose of BAY73-4506 in healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects between 18 and 45 years of age, inclusive
* BMI between 18 and 32 kg/m2 inclusive

Exclusion Criteria:

* Subjects with evidence of disease, conditions affecting drug absorption or metabolism
* Treatment with other investigational drug within 30 days
* History of regular alcohol or recreational drug consumption
* Use of prescription drugs within 14 days
* Use of nonprescription drugs and dietary supplement within 7 days
* Blood donation within 30 days

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2011-03; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve from zero to infinity ( Plasma AUCinf) of BAY73-4506 given alone or with ketoconazole. | 1 month
Peak plasma concentration (Cmax) of BAY73-4506 given alone or with ketoconazole | 1 month

SECONDARY OUTCOMES:
Plasma AUCinf of metabolites of a single oral dose BAY73-4506 given alone or with ketoconazole. | 1 month
Plasma Cmax of metabolites of a single oral dose BAY73-4506 given alone or with ketoconazole. | 1 month
Number of subjects with adverse events following a single oral dose of BAY73-4506, adminstered alone and concomitantly with ketoconazole. | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Brighton, Massachusetts, United States